CLINICAL TRIAL: NCT04136067
Title: A Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneous NNC0268-0965 in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Look at How Safe NNC0268-0965 is in People With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1965-4457; U1111-1227-8683 (Other: World Health Organization (WHO)); 2019-000754-58 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Intervention Model Description: 3 cohorts are planned. Each cohort will consist of 12 subjects, with 9 subjects being randomised to receive NNC0268-0965 and 3 subjects being randomised to insulin glargine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNC0268-0965 (Experimental): Participants will receive NNC0268-0965
  Interventions: Drug: NNC0268-0965
- Insulin glargine (Active Comparator): Participants will receive insulin glargine
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: NNC0268-0965 — One daily dose of 1.5, 4.0 or 6.0 nmol/kg administered s.c. (subcutaneously, under the skin) for 6 days
  Arms: NNC0268-0965
Drug: insulin glargine — One daily dose of 3.0 nmol/kg administered s.c. for 6 days
  Arms: Insulin glargine

SUMMARY:
This study looks at the safety and tolerability of the new medicine NNC0268-0965 (referred to as insulin 965), its concentration in the blood and its effect on the blood sugar for the treatment of diabetes. The study will test how insulin 965 is tolerated by the body, how it is taken up in the blood, how long it stays there and how the blood sugar is lowered. Participants will either get the new insulin 965 or the already marketed insulin glargine U100 (Lantus®) - which treatment is decided by chance. Participants will get six injections (one per day) of either insulin 965 or insulin glargine U100 under the skin of the left thigh. The study will last for about 5 weeks. Participants will have 6 clinic visits with the study doctor. Participants can only be in the study if the study doctor thinks that there are no risks for their health. Women can only take part in the study if they can't have children.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-64 years (both inclusive) at the time of signing informed consent.
* Diagnosed with type 2 diabetes mellitus 180 days or more prior to the day of screening.
* Male subject or female subject of non-child bearing potential. Non-child bearing potential being surgically sterilised (i.e. documented hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or being postmenopausal (as defined as no menses for 12 months without an alternative medical cause) prior to the day of screening.
* Current total daily insulin treatment between 0.25 (I)U/kg/day and 1.2 (I)U/kg/day (both inclusive).
* HbA1c equal to or below 9.5%

Exclusion Criteria:

* Male of reproductive age who, or whose partner(s), is not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice). Adequate contraceptive measures include that the male subject uses a condom during intercourse and that the partner practices adequate contraception (risk of pregnancy must be lower than 1%).
* Use of GLP-1 receptor agonists (e.g. exenatide, liraglutide, semaglutide) within 3 months prior to screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-08-23 (Actual); Study Completion 2020-08-23 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (AEs) | From IMP administration at day 1 (visit 2) until completion of post-treatment end-of-trial visit at day 12 (visit 5)
  Number of events

SECONDARY OUTCOMES:
Number of treatment-emergent hypoglycaemic episodes | From IMP administration at day 1 (visit 2) until completion of post-treatment end-of-trial visit at day 12 (visit 5)
  Number of episodes
Area under the serum NNC0268-0965 concentration-time curve during one dosing interval at steady state | From 0 to 24 hours after IMP administration at day 6 (visit 2)
  pmol*h/l
Maximum observed serum NNC0268-0965 concentration after the last dose | From 0 to 24 hours after IMP administration at day 6 (visit 2)
  pmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com